CLINICAL TRIAL: NCT06011941
Title: Safety and Feasibility of Modified Laparoscopic Transcystic Biliary Drainage in the Management of Cholecystocholedocholithiasis
Brief Title: Modified Laparoscopic Transcystic Biliary Drainage in the Management of Cholecystocholedocholithiasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81524
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Common Bile Duct Calculi; Acute; Cholecystitis, Choledocholithiasis; Acute Cholecystitis With Obstruction; Acute Cholangitis
MeSH Terms: conditions — Gallstones; Cholecystitis; Choledocholithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified laparoscopic transcystic biliary drainage (Experimental): A 7-Fr triple-lumen 30-cm central venous catheter was adopted to replace conventional 5-Fr ureteral catheter. Then we developed a continued suture and circling manner by the V-Loc closure device, which simultaneously covered and anchored the C-tube. Furthermore, the catheter was introduced through the abdominal wall located at 3 cm below the costal margin on the midaxillary line/the posterior axillary line, which was traditionally performed at the point below the midclavicular line on the right side.
  Interventions: Procedure: Modified laparoscopic transcystic biliary drainage

INTERVENTIONS:
Procedure: Modified laparoscopic transcystic biliary drainage — First, a needle was passed through a separate skin puncture wound 3 cm below the costal margin on the midaxillary line/posterior axillary line. Second, a lateral incision into the cystic duct was performed medially to allow insertion and embedding of the catheter. Third, a 7-Fr catheter was introduced through the abdominal wall via the cystic duct into the CBD. Fourth, if the position of the catheter inside the CBD was correct (the end of the tube reached the distal CBD but did not pass the papilla), the lateral incision of the cystic duct was closed by a V-Loc closure device using a single-layered, continuous suture in a circling manner to simultaneously cover and anchor the C-tube. After the procedure, an artificial fistula of 3 to 5 mm in length was formed.

SUMMARY:
The modified laparoscopic transcystic biliary drainage which we developed in the treatment of cholecystocholedocholithiasis has some advantages over conventional techniques.

Here, a 7-Fr triple-lumen 30-cm central venous catheter was adopted to replace conventional 5-Fr ureteral catheter, which extended the function of the C-tube.

Then we developed a continued suture and circling manner by the V-Loc closure device, which simultaneously covered and anchored the C-tube.

Theoretically, this modified laparoscopic transcystic drainage not only provide safe and effective bile duct drainage, but also provide a convenient access of treatment for postoperatively retained bile duct stones, which may expand the indication of initially laparoscopic operation in the management of cholecysto-choledocholithiasis.

DETAILED DESCRIPTION:
The modified laparoscopic transcystic biliary drainage which we developed in the treatment of cholecystocholedocholithiasis has some advantages over conventional techniques.

Here, a 7-Fr triple-lumen 30-cm central venous catheter was adopted (Arrow International Inc., Pennsylvania, U.S.A.) to replace conventional 5-Fr ureteral catheter, which extended the function of the C-tube.

Then we developed a continued suture and circling manner by the V-Loc closure device (Covidien V-Loc 180 3-0®, Mansfield, MA, US), which simultaneously covered and anchored the C-tube.

Furthermore, the catheter was introduced through the abdominal wall located at 3 cm below the costal margin on the midaxillary line/the posterior axillary line, which was traditionally performed at the point below the midclavicular line on the right side. Our modified path could avoid the compression of the C-tube by hepatic margin and hence decrease the dislocation of the C-tube. In addition, the retroperitoneal path may increase adherence development and sinus-tract formation.

More importantly, this path could easily be available when the patient be placed in the prone position for ERCP, which can conveniently facilitate the guidewire passed through the C-tube down to the duodenum to perform postoperative rendezvous technique.

Theoretically, this modified laparoscopic transcystic drainage not only provide safe and effective bile duct drainage, but also provide a convenient access of treatment for postoperatively retained bile duct stones, which may expand the indication of initially laparoscopic operation in the management of cholecysto-choledocholithiasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age;
* Patients with gallbladder stones and known or expected concomitant bile duct stones;
* Informed consent.

Exclusion Criteria:

* Biliary drainage is already present, e.g. preoperative ENBD, PTCD;
* Women who are pregnant;
* Declined consent;
* Inability to follow the procedures of the study, e.g. due to language problems and psychological disorders of the participant;
* Morbid obesity (BMI > 40);
* IV-VI class of the American Society of Anesthesiologists physical status classification;
* Contraindications for general anesthesia or surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
postoperative overall morbidity | 6 months
  All outcome variables will be assessed according to internationally accepted standards if available, that is, the consensus definitions for surgical and medical complications according to the Clavien-Dindo classification.
bile leakage | 6 months
  Bile leakage is determined according to the definition and grading of severity by the International Study Group of Liver Surgery.

SECONDARY OUTCOMES:
anchoring time of the C-tube | 6 months
  the consumption of time from needle puncture to ending of C-tube ligation
average daily drainage volume | 6 months
  the average volume of bile drainage per day
early dislodgement of C-tube | 6 months
  the dislodgement of C-tube before intended removal.

CONTACTS AND LOCATIONS:
Overall Officials: LINGFU ZHANG, Study Chair — 北京大学第三医院
Locations (1):
- Lingfu Zhang, Beijing, None Selected, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang LF, Hou CS, Xu Z, Wang LX, Ling XF, Wang G, Cui L, Xiu DR. [Clinical effect of laparoscopic transcystic drainage combined with common bile duct exploration for the patients with difficult biliary stones]. Beijing Da Xue Xue Bao Yi Xue Ban. 2022 Dec 18;54(6):1185-1189. doi: 10.19723/j.issn.1671-167X.2022.06.021. Chinese. PMID 36533353
- [Derived] Zhang YY, Wang G, Hou C, Xu Z, Wang L, Cui L, Ling X, Zhang L. Safety and effectiveness of modified laparoscopic transcystic biliary drainage in the treatment of choledocholithiasis: study protocol for a prospective single-arm clinical trial. BMJ Open. 2025 Apr 23;15(4):e089540. doi: 10.1136/bmjopen-2024-089540. PMID 40268483